CLINICAL TRIAL: NCT02606305
Title: A Phase 1b/2 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Mirvetuximab Soravtansine (IMGN853) in Combination With Bevacizumab, Carboplatin, Pegylated Liposomal Doxorubicin, Pembrolizumab, or Bevacizumab + Carboplatin, in Adults With Folate Receptor Alpha Positive Advanced Epithelial Ovarian Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer
Brief Title: Study of Mirvetuximab Soravtansine in Combination With Bevacizumab, Carboplatin, Pegylated Liposomal Doxorubicin, Pembrolizumab, or Bevacizumab + Carboplatin in Participants With Folate Receptor Alpha (FRα) Positive Advanced Epithelial Ovarian Cancer, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMGN853-0402; KEYNOTE PN409 (Other: Merck)
Record Dates: First submitted 2015-11-06; First posted 2015-11-17 (Estimated); Results first posted 2024-02-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Epithelial Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Epithelial ovarian cancer; Fallopian tube cancer; Primary peritoneal cancer; IMGN853; ADC; Antibody drug conjugate; ImmunoGen; Antibody; Phase 1; Folate receptor alpha; Mirvetuximab
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — mirvetuximab soravtansine; Bevacizumab; Carboplatin; liposomal doxorubicin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Regimen A (Mirvetuximab soravtansine + Bevacizumab) (Experimental): Mirvetuximab soravtansine + Bevacizumab administered on Day 1 of each 21-day cycle in Dose Escalation and Dose Expansion phase.
  Interventions: Drug: Mirvetuximab soravtansine; Drug: Bevacizumab
- Regimen B (Mirvetuximab soravtansine + Carboplatin) (Experimental): Mirvetuximab soravtansine + Carboplatin administered on Day 1 of each 21-day cycle in Dose Escalation phase.
  Interventions: Drug: Mirvetuximab soravtansine; Drug: Carboplatin
- Regimen C (Mirvetuximab soravtansine + Pegylated liposomal doxorubicin) (Experimental): Mirvetuximab soravtansine + Pegylated liposomal doxorubicin administered on Day 1 of each 28-day cycle in Dose Escalation Phase.
  Interventions: Drug: Mirvetuximab soravtansine; Drug: Pegylated Liposomal Doxorubicin
- Regimen D (Mirvetuximab soravtansine + Pembrolizumab) (Experimental): Mirvetuximab soravtansine + Pembrolizumab administered on Day 1 of each 21-day cycle in Dose Escalation and Dose Expansion phase.
  Interventions: Drug: Mirvetuximab soravtansine; Drug: Pembrolizumab
- Regimen E (Mirvetuximab soravtansine + Bevacizumab + Carboplatin) (Experimental): Mirvetuximab soravtansine + Bevacizumab + Carboplatin administered on Day 1 of each 21-day cycle in Dose Expansion phase.
  Interventions: Drug: Mirvetuximab soravtansine; Drug: Bevacizumab; Drug: Carboplatin

INTERVENTIONS:
Drug: Mirvetuximab soravtansine
  Other Names: IMGN853
Drug: Bevacizumab
  Arms: Regimen A (Mirvetuximab soravtansine + Bevacizumab); Regimen E (Mirvetuximab soravtansine + Bevacizumab + Carboplatin)
Drug: Carboplatin
  Arms: Regimen B (Mirvetuximab soravtansine + Carboplatin); Regimen E (Mirvetuximab soravtansine + Bevacizumab + Carboplatin)
Drug: Pegylated Liposomal Doxorubicin
  Arms: Regimen C (Mirvetuximab soravtansine + Pegylated liposomal doxorubicin)
Drug: Pembrolizumab
  Arms: Regimen D (Mirvetuximab soravtansine + Pembrolizumab)

SUMMARY:
This study comprises a Dose Escalation phase followed by a Dose Expansion phase. Dose Escalation part of the study will assess the safety and tolerability and determine the maximum tolerated dose (MTD) as the recommended Phase 2 (RP2D) dose for each regimen. Participants will be assigned to one of the 4 regimens in Dose Escalation phase: Regimen A: mirvetuximab soravtansine administered with bevacizumab; Regimen B: mirvetuximab soravtansine administered with carboplatin; Regimen C: mirvetuximab soravtansine administered with pegylated liposomal doxorubicin; or Regimen D: mirvetuximab soravtansine administered with pembrolizumab. Dose Expansion of the study will further assess safety, tolerability and preliminary anti-tumor activity of mirvetuximab soravtansine. A Dose Expansion phase is planned for Regimen A and Regimen D and will open pending Sponsor decision; participants enrolled in the Dose Expansion phase will receive study treatment at the MTD or RP2D determined during Dose Escalation. For Regimen A, participants in the Dose Expansion phase may be enrolled according to prior exposure to bevacizumab into 3 Dose Expansion Cohorts as follows: 1) Dose Expansion Cohort 1: bevacizumab naïve; 2) Dose Expansion Cohort 2: bevacizumab pretreated; and 3) Dose Expansion Cohort 3: one to three prior treatments, one of which could have been bevacizumab. A triplet Regimen (Regimen E: mirvetuximab soravtansine + bevacizumab + carboplatin) will be opened to evaluate the safety and tolerability and to assess any early signs of activity in participants dosed with the combination regimen. All mirvetuximab soravtansine doses were calculated according to adjusted ideal body weight.

DETAILED DESCRIPTION:
Participants will continue to receive mirvetuximab soravtansine and/or the combination agent until progressive disease (PD), unacceptable toxicity, or withdrawal of consent, whichever comes first, or until the Sponsor terminates the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with advanced epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer
* Folate receptor α (FRα) positive tumor expression as defined in the protocol
* Willing to provide an archival tumor tissue block or slides or undergo tumor biopsy. New tumor biopsy (Cycle 2 Day 8) is required for Regimen D.
* Measurable disease

Exclusion Criteria:

* Primary platinum-refractory disease
* Diagnosis of clear cell, low grade ovarian cancer or mixed tumors
* Serious concurrent illness or clinically relevant active infection, including but not limited to known diagnosis of human immunodeficiency virus (HIV) and hepatitis B or C, as defined in the protocol
* Active autoimmune disease requiring systemic therapy in past 2 years (for Regimen D only)
* Women who are pregnant or breastfeeding
* Male participants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - University of California at Los Angeles, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - City of Hope, Reno, Nevada
  - The Ohio State University, Hilliard, Ohio
  - Peggy and Charles Stephenson Oklahoma Cancer Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Universitaire Ziekenhuizen (UZ) Leuven - Gasthuisberg - Leuvens Kankerinstituut, Leuven, Belgium
- Canada (2):
  - Centre Hospitalier de l'universite de Montreal (CHUM), Montreal
  - McGill University Health Center, Montreal
- Spain (2):
  - Hospital Vall D'Hebron, Barcelona
  - MD Anderson, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg: Participants were administered mirvetuximab soravtansine 5 milligrams (mg)/kilograms (kg) + bevacizumab 15 mg/kg on Day 1 of each 21-day cycle.
- Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg: Participants were administered mirvetuximab soravtansine 6 mg/kg + bevacizumab 15 mg/kg on Day 1 of each 21-day cycle.
- Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve: Participants not previously treated with bevacizumab (bevacizumab naïve) were administered mirvetuximab soravtansine 6 mg/kg + bevacizumab 15 mg/kg on Day 1 of each 21-day cycle.
- Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated: Participants who were pre-treated with bevacizumab were administered mirvetuximab soravtansine 6 mg/kg + bevacizumab 15 mg/kg on Day 1 of each 21-day cycle.
- Regimen A Dose Expansion Cohort 3: Pt-agnostic:: Participants with at least 1 but no more than 3 prior systemic treatment regimens, where prior regimens may have included bevacizumab were administered mirvetuximab soravtansine 6 mg/kg + bevacizumab 15 mg/kg.
- Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4: Participants were administered mirvetuximab soravtansine 5 mg/kg + carboplatin area under the time-concentration curve (AUC4) on Day 1 of each 21-day cycle.
- Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5: Participants were administered mirvetuximab soravtansine 5 mg/kg + carboplatin AUC5 on Day 1 of each 21-day cycle.
- Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5: Participants were administered mirvetuximab soravtansine 6 mg/kg + carboplatin AUC5 on Day 1 of each 21-day cycle.
- Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2: Participants were administered mirvetuximab soravtansine 5 mg/kg + pegylated liposomal doxorubicin (PLD) 30 mg/meter squared (m^2) on Day 1 of each 28-day cycle.
- Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2: Participants were administered mirvetuximab soravtansine 5 mg/kg + PLD 40 mg/m^2 on Day 1 of each 28-day cycle.
- Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2: Participants were administered mirvetuximab soravtansine 6 mg/kg + PLD 40 mg/m^2 on Day 1 of each 28-day cycle.
- Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg: Participants were administered mirvetuximab soravtansine 5 mg/kg + pembrolizumab 200 mg on Day 1 of each 21-day cycle.
- Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg; Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg: Participants were administered mirvetuximab soravtansine 6 mg/kg + pembrolizumab 200 mg on Day 1 of each 21-day cycle.
- Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin: Participants were administered mirvetuximab soravtansine 6 mg/kg + bevacizumab 15 mg/kg + carboplatin AUC5 on Day 1 of each 21-day cycle.
Period: Dose Escalation: Regimens A, B, C and D
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Started | 3 | 11 | 0 | 0 | 0 | 4 | 4 | 10 | 4 | 5 | 7 | 4 | 10 | 0 | 0
Received at Least 1 Dose of Study Drug | 3 | 11 | 0 | 0 | 0 | 4 | 4 | 10 | 4 | 5 | 7 | 4 | 10 | 0 | 0
Completed | 3 | 11 | 0 | 0 | 0 | 4 | 4 | 10 | 4 | 5 | 7 | 4 | 10 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion: Regimens A and D
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Started | 0 | 0 | 21 | 34 | 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 46 | 0
Received at Least 1 Dose of Study Drug | 0 | 0 | 21 | 34 | 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 21 | 34 | 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 46 | 0
Period: Triplet Dose: Regimen E
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg: Participants were administered mirvetuximab soravtansine 5 mg/kg + bevacizumab 15 mg/kg on Day 1 of each 21-day cycle.
- Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4: Participants were administered mirvetuximab soravtansine 5 mg/kg + carboplatin AUC4 on Day 1 of each 21-day cycle.
- Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2: Participants were administered mirvetuximab soravtansine 5 mg/kg + PLD 30 mg/m^2 on Day 1 of each 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin | Total
Number analyzed (Participants) | 3 | 11 | 21 | 34 | 60 | 4 | 4 | 10 | 4 | 5 | 7 | 4 | 10 | 46 | 41 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (11.85) | 65.5 (8.43) | 62.2 (7.40) | 61.4 (9.99) | 61.4 (9.87) | 59.3 (9.14) | 67.0 (7.07) | 66.0 (10.33) | 59.5 (12.07) | 65.2 (4.66) | 60.6 (5.35) | 58.3 (6.18) | 63.5 (10.81) | 61.1 (8.64) | 63.8 (9.40) | 62.3 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 21 | 34 | 60 | 4 | 4 | 10 | 4 | 5 | 7 | 4 | 10 | 46 | 41 | 264
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 6
  Not Hispanic or Latino | 3 | 11 | 21 | 32 | 58 | 4 | 4 | 9 | 4 | 4 | 7 | 4 | 10 | 45 | 39 | 255
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  White | 3 | 10 | 21 | 32 | 53 | 4 | 4 | 10 | 4 | 5 | 7 | 4 | 10 | 43 | 39 | 249
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse events (AEs) were any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function that developed or worsened during the clinical study, not necessarily having a causal relationship to study drug. Severity was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening, Grade 5=death. Serious AEs included death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes previously listed. TEAEs were any AE that emerged on or after the first dose, and within 30 days of the last dose. Serious and other non-serious AEs regardless of causality are reported in the AE module.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (maximum exposure: 238.3 weeks)
Population: All participants who were enrolled and received at least 1 dose of study drug. Data were reported by dose group and where applicable the dose-escalation and expansion phases were combined to report data by dose group.
Measure: Count of Participants; unit: Participants
Groups:
- Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg: Participants were administered mirvetuximab soravtansine 5 mg/kg + bevacizumab 15 mg/kg on Day 1 of each 21-day cycle.
- Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg: All participants who were administered mirvetuximab soravtansine 6 mg/kg + bevacizumab 15 mg/kg on Day 1 of each 21-day cycle in the dose escalation and dose expansion phases.
- Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4: Participants were administered mirvetuximab soravtansine 5 mg/kg + carboplatin AUC4 on Day 1 of each 21-day cycle.
- Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5: Participants were administered mirvetuximab soravtansine 5 mg/kg + carboplatin AUC5 on Day 1 of each 21-day cycle.
- Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5: Participants were administered mirvetuximab soravtansine 6 mg/kg + carboplatin AUC5 on Day 1 of each 21-day cycle.
- Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2: Participants were administered mirvetuximab soravtansine 5 mg/kg + PLD 30 mg/m^2 on Day 1 of each 28-day cycle.
- Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2: Participants were administered mirvetuximab soravtansine 5 mg/kg + PLD 40 mg/m^2 administered on Day 1 of each 28-day cycle.
- Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2: Participants were administered mirvetuximab soravtansine 6 mg/kg + PLD 40 mg/m^2 on Day 1 of each 28-day cycle.
- Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg: Participants were administered mirvetuximab soravtansine 5 mg/kg + pembrolizumab 200 mg on Day 1 of each 21-day cycle.
- Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg: All participants who were administered mirvetuximab soravtansine 6 mg/kg + pembrolizumab 200 mg on Day 1 of each 21-day cycle in the dose escalation and dose expansion phases.
- Mirvetuximab Soravtansine + Bevacizumab + Carboplatin: Participants were administered mirvetuximab soravtansine 6 mg/kg + bevacizumab 15 mg/kg + carboplatin AUC5 on Day 1 of each 21-day cycle.
Arm/Group | Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 3 | 126 | 4 | 4 | 10 | 4 | 5 | 7 | 4 | 56 | 41
Participants
  Any TEAE | 3 | 126 | 4 | 4 | 10 | 4 | 4 | 7 | 4 | 56 | 41
  SAEs | 2 | 49 | 2 | 4 | 3 | 1 | 2 | 3 | 2 | 25 | 17
  Grade >=3 TEAEs | 2 | 85 | 2 | 4 | 7 | 2 | 3 | 6 | 1 | 30 | 37

2. Primary Outcome: Dose Expansion (Regimens A and D) and Triplet (Regimen E): Objective Response Rate (ORR); Percentage of Participants With Confirmed Response, as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: ORR was defined as percentage of participants with confirmed response (complete response [CR] + partial response [PR]). CR: Disappearance of all target or non-target lesions. All pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR: At least 30 percent (%) decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline SLD. The 95% confidence interval (CI) was based on binomial distribution.
Time Frame: From first dose of study drug until first CR or PR (maximum exposure: 238.3 weeks)
Population: Response-Evaluable Population: All participants who received at least 1 dose of study treatment, had radiographic assessment at baseline received at least 1 dose of combination treatment, and at least 1 post-dose radiographic tumor assessment or have died within 105 days of first dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 21 | 34 | 60 | 45 | 41
percentage of participants | 52 [29.78 to 74.29] | 29 [15.10 to 47.48] | 50 [36.81 to 63.19] | 27 [14.60 to 41.94] | 83 [67.94 to 92.85]

3. Secondary Outcome: Dose Escalation (Regimens A Through D): ORR; Percentage of Participants With Confirmed Response, as Assessed by RECIST Version 1.1
Description: ORR was defined as percentage of participants with confirmed response (CR + PR). CR: Disappearance of all target or non-target lesions. All pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least 30% decrease in the SLD of target lesions, taking as reference the baseline SLD.
Time Frame: From first dose of study drug until first CR or PR (maximum exposure: 238.3 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2: Participants were administered mirvetuximab soravtansine 6 mg/kg + PLD 40 mg/m^2 administered on Day 1 of each 28-day cycle.
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 3 | 11 | 4 | 4 | 9 | 4 | 5 | 7 | 4 | 10
percentage of participants | 0 [0.00 to 0.00] | 45 [16.75 to 76.62] | 50 [6.76 to 93.24] | 50 [6.76 to 93.24] | 89 [51.75 to 99.72] | 0 [0.00 to 0.00] | 20 [0.51 to 71.64] | 29 [3.67 to 70.96] | 25 [0.63 to 80.59] | 50 [18.71 to 81.29]

4. Secondary Outcome: Progression-Free Survival (PFS); Time From the Date Of First Dose Until The Date Of Progressive Disease (PD) Or Death By Any Cause, As Defined By RECIST Version 1.1
Description: PFS was defined as the time from the date of the first dose of study drug until the date of PD or death from any cause, whichever occurred first, estimated using the Kaplan-Meier method. PFS was defined based on radiological assessments and determined by the investigator. PD was defined as at least a 20% increase in the SLD of target lesions, taking as reference the smallest (nadir) SLD since and including baseline. In addition to the relative increase of 20%, the SLD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions and appearance of new lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: From first dose of study drug until the date of PD or death by any cause (maximum exposure: 238.3 weeks)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg: Participants were administered mirvetuximab soravtansine 6 mg/kg + bevacizumab 15 mg/kg administered on Day 1 of each 21-day cycle.
- Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2: Participants were administered mirvetuximab soravtansine 5 mg/kg + PLD 40 mg/m^2 administered on Day 1 of each 28-day cycle.
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 3 | 11 | 21 | 34 | 60 | 4 | 4 | 9 | 4 | 5 | 7 | 4 | 10 | 45 | 41
months | 13.49 [11.76 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 8.80 [1.18 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 9.92 [7.13 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 6.77 [4.63 to 10.71] | 8.28 [6.34 to 11.01] | 13.52 [10.38 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 32.94 [10.38 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 16.46 [6.97 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | NA [1.68 to NA] — Due to smaller number of events, median and upper 95% CI could not be calculated. | 7.03 [0.26 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 7.23 [1.45 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 2.53 [1.18 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 9.46 [1.38 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 4.17 [2.79 to 5.52] | 13.50 [9.86 to 16.30]

5. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1 by Investigator Assessment
Description: DOR was defined as the time from the date of the first response (CR or PR), to the date of PD or death from any cause, whichever occurred first. DOR was only defined for patients who had a best overall response of CR or PR, estimated using the Kaplan-Meier method. The response-evaluable population included all patients with radiographic assessment at baseline, who received at least 1 dose of combination treatment and had at least 1 post-dose radiographic tumor assessment or who died within 105 days of first dose.
Time Frame: From the date of first objective response to the time of PD (maximum exposure: 238.3 weeks)
Population: Response-Evaluable Population: All participants who received at least 1 dose of study treatment, had radiographic assessment at baseline received at least 1 dose of combination treatment, and at least 1 post-dose radiographic tumor assessment or have died within 105 days of first dose. Only participants who had best overall response of CR or PR were analyzable.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5: Participants were administered mirvetuximab soravtansine 6 mg/kg + carboplatin AUC5 administered on Day 1 of each 21-day cycle.
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 0 | 5 | 11 | 10 | 30 | 2 | 2 | 8 | 0 | 1 | 2 | 1 | 5 | 12 | 34
months |  | NA [2.76 to NA] — Due to smaller number of events, median and upper 95% CI could not be calculated. | 11.96 [2.99 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 14.06 [3.91 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 10.38 [6.93 to 13.67] | NA [6.05 to NA] — Due to smaller number of events, median and upper 95% CI could not be calculated. | 31.77 [9.20 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 12.12 [4.40 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. |  | NA [NA to NA] — Due to smaller number of events, median and upper 95% CI could not be calculated. | NA [5.29 to NA] — Due to smaller number of events, median and upper 95% CI could not be calculated. | 3.42 [NA to NA] — Due to smaller number of events, 95% CI could not be calculated. | 8.31 [6.93 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 4.37 [2.79 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 10.87 [8.71 to 15.15]

6. Secondary Outcome: Gynecologic Cancer Intergroup (GCIG) Cancer Antigen (CA)-125 Clinical Response Rate by Investigator Assessment
Description: A CA-125 response was defined as a ≥ 50% reduction in CA-125 levels from baseline. GCIG CA125 response rate was defined as the number of participants with a CA-125 confirmed response divided by the number of participants in the CA-125 response-evaluable population multiplied by 100. The CA-125 evaluable population included all participants whose pretreatment sample was ≥2.0 times the upper limit of normal, within 2 weeks prior to the first dose of combination treatment, and who had at least 1 post-baseline CA-125 evaluation.
Time Frame: From first dose of study drug until first CR or PR (maximum exposure: 238.3 weeks)
Population: CA125 Evaluable Population: All participants whose pretreatment sample is ≥ 2.0 times the upper limit of normal (ULN), within 2 weeks prior to the first dose of combination treatment, and who have at least 1 post-baseline CA125 evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 1 | 10 | 16 | 26 | 56 | 3 | 3 | 7 | 3 | 2 | 6 | 2 | 8 | 37 | 27
percentage of participants | 100 [2.5 to 100.0] | 60 [26.2 to 87.8] | 75 [47.6 to 92.7] | 65 [44.3 to 82.8] | 71 [57.8 to 82.7] | 67 [9.4 to 99.2] | 100 [29.2 to 100.0] | 86 [42.1 to 99.6] | 0 [NA to NA] — Due to no events, 95% CI could not be calculated. | 50 [1.3 to 98.7] | 50 [11.8 to 88.2] | 0 [NA to NA] — Due to no events, 95% CI could not be calculated. | 63 [24.5 to 91.5] | 46 [29.5 to 63.1] | 100 [87.2 to 100.0]

7. Secondary Outcome: Pharmacokinetics (PK) Parameter: Maximum Plasma Concentration (Cmax) of Mirvetuximab Soravtansine and Total Antibody
Description: Blood samples from participants were analyzed to characterize the PK of mirvetuximab soravtansine when administered in 3- or 4-week cycles. Results are reported in micrograms/milliliter (µg/mL).
Time Frame: Cycles 1 and 3: Day 1 (pre-infusion, within 10 minutes of end of infusion [EOI], and 6 hours post-infusion); Days 2 and 3 (24- and 48-hours post-infusion); Days 8 and 15 (additionally at Day 22 for Regimen C)
Population: Response-Evaluable Population: All participants who received at least 1 dose of study treatment, had radiographic assessment at baseline received at least 1 dose of combination treatment, and at least 1 post-dose radiographic tumor assessment or have died within 105 days of first dose. The 'Number Analyzed' signifies participants evaluable for the specified categories.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg: Participants were administered mirvetuximab soravtansine 6 mg/kg + pembrolizumab 200 mg administered on Day 1 of each 21-day cycle.
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 3 | 11 | 20 | 34 | 60 | 4 | 4 | 10 | 4 | 5 | 7 | 4 | 10 | 46 | 41
µg/mL
  Mirvetuximab Soravtansine: Cycle 1 | 135 (9.2) | 137 (14.5) | 159 (30.4) | 159 (17.2) | 150 (17.2) | 118 (15.4) | 108 (15.7) | 144 (19.3) | 115 (21.5) | 114 (15.8) | 146 (16.8) | 112 (4) | 156 (13.2) | 151 (17.4) | 144 (18.5)
  Mirvetuximab Soravtansine: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 58 | 4 | 4 | 9 | 2 | 4 | 7 | 3 | 8 | 41 | 41
  Mirvetuximab Soravtansine: Cycle 3 | NA (NA) — Geometric mean Cmax could not be calculated for n<3 | 148 (15.8) | 164 (12.4) | 174 (14.1) | 137 (144) | 46 (999) | 121 (15.1) | 147 (12.1) | NA (NA) — Geometric mean Cmax could not be calculated for n<3 | 137 (15.4) | 142 (6.03) | 114 (20) | 165 (10.6) | 159 (15.7) | 128 (66.1)
  Total Antibody: Cycle 1 | 121 (11.8) | 122 (12.9) | 152 (31.1) | 148 (24.2) | 153 (13) | 118 (18.2) | 102 (16.4) | 129 (11.8) | 111 (23.5) | 114 (18.6) | 152 (17.2) | 94.7 (34.2) | 124 (11.8) | 146 (16.4) | 144 (18.3)
  Total Antibody: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 58 | 4 | 4 | 10 | 2 | 4 | 7 | 3 | 8 | 41 | 41
  Total Antibody: Cycle 3 | NA (NA) — Geometric mean Cmax could not be calculated for n<3 | 147 (25.1) | 177 (26.6) | 175 (22.7) | 180 (41) | 57.9 (238) | 122 (20.9) | 149 (15.5) | NA (NA) — Geometric mean Cmax could not be calculated for n<3 | 124 (3.32) | 140 (19) | 114 (17.8) | 160 (23) | 165 (17.4) | 146 (44.2)

8. Secondary Outcome: PK Parameter: Cmax of N2'-[4-[(3-carboxypropyl)Dithio]-4-methyl-1-oxo-2-sulfopentyl]-N2'-Deacetylmaytansine (DM4) and S-methyl DM4 (SmDM4)
Description: Blood samples from participants were analyzed to characterize the PK of mirvetuximab soravtansine when administered in 3- or 4-week cycles. Results are reported in nanograms (ng)/mL.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 3 | 11 | 20 | 35 | 60 | 4 | 4 | 10 | 4 | 5 | 7 | 4 | 10 | 46 | 41
ng/mL
  DM4: Cycle 1 | 3.04 (21.8) | 4.71 (32.9) | 5.51 (35.8) | 6.32 (33.8) | 5.59 (37.5) | 2.96 (8.85) | 3.72 (28.7) | 6.4 (27.7) | 4.12 (47.5) | 3.93 (18.3) | 6.58 (86.4) | 4.54 (49.3) | 5.6 (31.2) | 5.27 (35.3) | 4.52 (38.4)
  DM4: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 58 | 4 | 4 | 9 | 2 | 4 | 7 | 3 | 8 | 41 | 41
  DM4: Cycle 3 | NA (NA) — Geometric mean Cmax could not be calculated for n<3 | 5.06 (30.5) | 4.57 (27.3) | 6.16 (43.8) | 5.45 (69.1) | 3.06 (23.4) | 3.38 (15) | 5.66 (31.2) | NA (NA) — Geometric mean Cmax could not be calculated for n<3 | 5.1 (34.4) | 7.02 (70.8) | 3.91 (5.81) | 4.91 (37.3) | 4.95 (33.3) | 4.44 (25.7)
  S-methyl DM4: Cycle 1 | 3.61 (26.7) | 9.6 (65.5) | 11.5 (61.7) | 12.2 (68.9) | 12.2 (62.6) | 5.75 (56.3) | 7.91 (46.9) | 13 (37.5) | 7.23 (50.8) | 7.51 (58.1) | 11.9 (77.1) | 11.3 (56.6) | 17 (91.8) | 12.8 (63.6) | 8.64 (71.7)
  S-methyl DM4: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 58 | 4 | 4 | 9 | 2 | 4 | 7 | 3 | 8 | 41 | 41
  S-methyl DM4: Cycle 3 | NA (NA) — Geometric mean Cmax could not be calculated for n<3 | 12.3 (71.1) | 11.8 (55.7) | 12.2 (51.9) | 12.5 (89.2) | 3.21 (220) | 6.79 (59.1) | 14.1 (43.9) | NA (NA) — Geometric mean Cmax could not be calculated for n<3 | 10.8 (55.7) | 17.6 (63) | 16.2 (11.1) | 18 (52.9) | 13 (71.6) | 9.49 (104)

9. Secondary Outcome: PK Parameter: Area Under the Time-Concentration Curve From Time 0 To Infinite Time (AUCinf) of Mirvetuximab Soravtansine and Total Antibody
Description: Blood samples from participants were analyzed to characterize the PK of mirvetuximab soravtansine when administered in 3- or 4-week cycles. Results are reported in mg*hours (h)/mL.
Time Frame: Cycles 1 and 3: Day 1 (pre-infusion, within 10 minutes of EOI, and 6 hours post-infusion); Days 2 and 3 (24- and 48-hours post-infusion); Days 8 and 15 (additionally at Day 22 for Regimen C)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/mL
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 3 | 11 | 20 | 34 | 60 | 4 | 4 | 10 | 4 | 4 | 7 | 4 | 10 | 45 | 41
mg*h/mL
  Mirvetuximab Soravtansine: Cycle 1 | 16.1 (2.34) | 17 (13.9) | 18.6 (22.2) | 18.4 (22.1) | 17.5 (19.8) | 14.8 (13.8) | 11.3 (23) | 16.3 (26.7) | 14 (23.8) | 15.2 (34.1) | 16.2 (33.1) | 12.1 (19.1) | 17 (30.5) | 16.9 (32.9) | 17.8 (26.3)
  Mirvetuximab Soravtansine: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 53 | 3 | 4 | 8 | 2 | 4 | 7 | 3 | 8 | 40 | 39
  Mirvetuximab Soravtansine: Cycle 3 | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 21.6 (37.2) | 22.7 (14.1) | 22.8 (24.9) | 22.3 (16.7) | 15.2 (22.1) | 17.9 (16.1) | 19.9 (26.5) | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 17.4 (19.4) | 16.4 (14.1) | 14.4 (32.1) | 20.2 (28.2) | 20.9 (30.8) | 19.7 (20)
  Total Antibody: Cycle 1: number analyzed (Participants) | 2 | 7 | 15 | 20 | 50 | 4 | 4 | 9 | 4 | 3 | 6 | 4 | 7 | 31 | 32
  Total Antibody: Cycle 1 | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 20.6 (22.2) | 24.5 (31.4) | 23.5 (34.2) | 25.8 (22) | 18 (22.2) | 13.3 (29) | 21.6 (35.1) | 20.1 (55) | 17.8 (73.5) | 24.8 (26.2) | 16.8 (16.3) | 18.4 (49.1) | 20 (44.6) | 25 (25.4)
  Total Antibody: Cycle 3: number analyzed (Participants) | 2 | 4 | 10 | 18 | 28 | 2 | 0 | 3 | 2 | 2 | 6 | 2 | 3 | 20 | 17
  Total Antibody: Cycle 3 | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 24.2 (31.3) | 36.1 (23) | 34.7 (49.3) | 39.2 (20.1) | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 |  | 30 (26) | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 29.1 (33.6) | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 20.1 (29.7) | 28.9 (55.2) | 35.8 (32.6)

10. Secondary Outcome: PK Parameter: AUCinf of Intact DM4 and SmDM4
Description: Blood samples from participants were analyzed to characterize the PK of mirvetuximab soravtansine when administered in 3- or 4-week cycles. Note that '9999' is used because AUCinf cannot be calculated for n<3.
Time Frame: as for outcome 9
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 2 | 10 | 20 | 32 | 57 | 4 | 4 | 9 | 4 | 4 | 7 | 4 | 10 | 46 | 37
ng*h/mL
  DM4: Cycle 1: number analyzed (Participants) | 2 | 10 | 20 | 29 | 54 | 4 | 4 | 9 | 3 | 4 | 5 | 3 | 10 | 43 | 37
  DM4: Cycle 1 | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 249 (12.6) | 253 (28.2) | 289 (30.9) | 272 (28.4) | 161 (15.2) | 202 (21.6) | 315 (55.6) | 223 (64.8) | 180 (19.7) | 262 (49.6) | 192 (33.2) | 269 (17.7) | 261 (31.6) | 256 (40.7)
  DM4: Cycle 3: number analyzed (Participants) | 2 | 8 | 15 | 29 | 50 | 3 | 4 | 8 | 1 | 3 | 6 | 3 | 8 | 39 | 36
  DM4: Cycle 3 | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 282 (14.1) | 263 (31.4) | 315 (36.5) | 285 (27.2) | 146 (22) | 180 (17.4) | 295 (31.3) | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 200 (24.2) | 289 (53.6) | 163 (7.42) | 245 (29.7) | 260 (38.2) | 243 (29.2)
  S-methyl DM4: Cycle 1: number analyzed (Participants) | 2 | 8 | 19 | 32 | 57 | 3 | 2 | 9 | 4 | 4 | 6 | 4 | 9 | 40 | 35
  S-methyl DM4: Cycle 1 | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 1700 (51.5) | 1710 (73.2) | 1980 (60.7) | 2120 (62.1) | 1370 (49.2) | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 2160 (56.5) | 1510 (63.7) | 1660 (119) | 1830 (72.2) | 2050 (50) | 2930 (91.3) | 2460 (70.8) | 1830 (61.2)
  S-methyl DM4: Cycle 3: number analyzed (Participants) | 2 | 10 | 17 | 31 | 50 | 3 | 3 | 8 | 2 | 4 | 7 | 2 | 8 | 38 | 36
  S-methyl DM4: Cycle 3 | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 1730 (76.3) | 1620 (58.5) | 1930 (52.9) | 2120 (57.8) | 1130 (14.3) | 1600 (49.6) | 1600 (52.4) | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 1800 (80.8) | 2290 (70) | NA (NA) — Geometric mean AUCinf could not be calculated for n<3 | 2280 (61.9) | 2080 (75.5) | 1550 (61.8)

11. Secondary Outcome: PK Parameter: Terminal Half-Life (t½) of Mirvetuximab Soravtansine, Total Antibody, DM4, and SmDM4
Description: Blood samples from participants were analyzed to characterize the PK of mirvetuximab soravtansine when administered in 3- or 4-week cycles. PK parameters were calculated using standard non-compartmental methods.
  The terminal t½ is an estimate (extrapolation) of the time it takes for the concentration or amount in the body of that drug to be reduced by exactly one-half (50%). If extrapolated AUC was greater than 20% (due to insufficient number of participants with data samples) the upper range of t½ was not reported.
Time Frame: Cycles 1 and 3: Day 1 (pre-infusion, within 10 minutes of EOI, and 6 hours post-infusion); Days 2 and 3 (24- and 48-hours post-infusion); Days 8 and 15 (up to 336 hours) (additionally at Day 22 for Regimen C)
Population: as for outcome 7
Measure: Median (Full Range); unit: h
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 3 | 11 | 20 | 34 | 60 | 4 | 4 | 10 | 4 | 4 | 7 | 4 | 10 | 46 | 41
h
  Mirvetuximab Soravtansine: Cycle 1 | 104 [104 to 143] | 123 [89.5 to 146] | 124 [76 to 154] | 121 [59.1 to 161] | 126 [82.1 to 168] | 117 [97.8 to 119] | 123 [97.7 to 152] | 128 [92.5 to 151] | 124 [114 to 176] | 148 [67.6 to 187] | 137 [86.2 to 156] | 120 [115 to 135] | 126 [70.3 to 184] | 126 [57.5 to 173] | 122 [85.9 to 172]
  Mirvetuximab Soravtansine: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 54 | 3 | 4 | 9 | 2 | 4 | 7 | 3 | 8 | 41 | 40
  Mirvetuximab Soravtansine: Cycle 3 | NA [NA to NA] — As per the PK analysis plan, t½ statistics were not calculated when less than 3 individual values were available. | 132 [93.7 to 157] | 132 [100 to 178] | 128 [65.9 to 181] | 130 [84.9 to 199] | 124 [119 to 146] | 124 [116 to 161] | 137 [108 to 165] | NA [NA to NA] — As per the PK analysis plan, t½ statistics were not calculated when less than 3 individual values were available. | 175 [76.6 to 237] | 119 [103 to 140] | 114 [97.8 to 118] | 132 [99.9 to 173] | 133 [62.5 to 192] | 140 [97.6 to 202]
  Total Antibody: Cycle 1 | 142 [107 to 226] | 206 [114 to 330] | 182 [87.9 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 221 [76.2 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 200 [119 to 315] | 189 [156 to 225] | 170 [165 to 286] | 208 [109 to 333] | 231 [200 to 299] | 282 [80.6 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 249 [182 to 314] | 184 [168 to 209] | 182 [68.9 to 269] | 196 [58 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 215 [111 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported.
  Total Antibody: Cycle 3: number analyzed (Participants) | 2 | 9 | 18 | 32 | 54 | 3 | 4 | 9 | 2 | 4 | 7 | 3 | 8 | 41 | 41
  Total Antibody: Cycle 3 | NA [NA to NA] — As per the PK analysis plan, t½ statistics were not calculated when less than 3 individual values were available. | 235 [165 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 214 [127 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 228 [86.8 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 216 [146 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 214 [143 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 290 [160 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 214 [163 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | NA [NA to NA] — As per the PK analysis plan, t½ statistics were not calculated when less than 3 individual values were available. | 337 [94.5 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 230 [88.4 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 197 [135 to 278] | 269 [170 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 232 [70.3 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 251 [148 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported.
  DM4: Cycle 1: number analyzed (Participants) | 3 | 10 | 20 | 30 | 55 | 4 | 4 | 9 | 4 | 4 | 5 | 3 | 10 | 45 | 39
  DM4: Cycle 1 | 49.9 [40.5 to 121] | 74.4 [47.8 to 104] | 70.2 [47.2 to 99.7] | 61.9 [43.9 to 100] | 63.9 [40.1 to 124] | 59.4 [45 to 73.3] | 60.6 [40.4 to 124] | 52.4 [39.6 to 115] | 65.9 [48.6 to 120] | 55.8 [51.7 to 65.6] | 57.4 [43 to 91.4] | 46.4 [38 to 62.9] | 73.6 [42.8 to 131] | 59.4 [29.8 to 219] | 57.5 [39.9 to 116]
  DM4: Cycle 3: number analyzed (Participants) | 2 | 8 | 17 | 30 | 51 | 3 | 4 | 9 | 1 | 3 | 7 | 3 | 8 | 39 | 37
  DM4: Cycle 3 | NA [NA to NA] — As per the PK analysis plan, t½ statistics were not calculated when less than 3 individual values were available. | 83.8 [40.8 to 94.1] | 73.9 [32.8 to 102] | 71.1 [39.4 to 111] | 78.3 [19.1 to 109] | 68 [52.3 to 69.6] | 63.6 [59 to 111] | 74.1 [52.7 to 101] | NA [NA to NA] — As per the PK analysis plan, t½ statistics were not calculated when less than 3 individual values were available. | 96 [71.7 to 105] | 64.4 [45.5 to 115] | 46.5 [41.7 to 65.5] | 64.6 [53.3 to 109] | 64 [33 to 161] | 63 [45.2 to 109]
  S-methyl DM4: Cycle 1: number analyzed (Participants) | 2 | 8 | 20 | 32 | 58 | 3 | 2 | 9 | 4 | 4 | 7 | 4 | 9 | 41 | 38
  S-methyl DM4: Cycle 1 | NA [NA to NA] — As per the PK analysis plan, t½ statistics were not calculated when less than 3 individual values were available. | 132 [97 to 178] | 126 [97.8 to 245] | 129 [81.7 to 217] | 139 [94.1 to 209] | 128 [96 to 151] | NA [NA to NA] — As per the PK analysis plan, t½ statistics were not calculated when less than 3 individual values were available. | 132 [99.2 to 165] | 168 [133 to 220] | 181 [156 to 285] | 154 [126 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of t½ upper range, therefore, not reported. | 132 [106 to 169] | 134 [104 to 163] | 127 [73.4 to 253] | 126 [84.4 to 292]
  S-methyl DM4: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 31 | 50 | 3 | 4 | 10 | 2 | 4 | 7 | 3 | 8 | 41 | 37
  S-methyl DM4: Cycle 3 | NA [NA to NA] — As per the PK analysis plan, t½ statistics were not calculated when less than 3 individual values were available. | 128 [97.3 to 216] | 132 [94.8 to 172] | 126 [86.7 to 207] | 121 [79.1 to 196] | 140 [127 to 186] | 168 [107 to 233] | 124 [100 to 155] | NA [NA to NA] — As per the PK analysis plan, t½ statistics were not calculated when less than 3 individual values were available. | 182 [165 to 251] | 169 [105 to 213] | 171 [130 to 192] | 148 [120 to 158] | 140 [88.3 to 253] | 138 [84.9 to 275]

12. Secondary Outcome: PK Parameter: Clearance (CL) of Mirvetuximab Soravtansine and Total Antibody
Description: Blood samples from participants were analyzed to characterize the PK of mirvetuximab soravtansine when administered in 3- or 4-week cycles.
Time Frame: as for outcome 9
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 3 | 11 | 20 | 34 | 60 | 4 | 4 | 10 | 4 | 4 | 7 | 4 | 10 | 45 | 41
mL/h
  Mirvetuximab Soravtansine: Cycle 1 | 19.2 (18.8) | 22 (17.2) | 22 (29.1) | 20.9 (23.3) | 23.4 (23.8) | 19.9 (10.1) | 28.9 (17) | 22 (26.1) | 21.2 (22.3) | 23.3 (38.6) | 24.5 (41.3) | 29.2 (17.1) | 23.9 (34.5) | 22.8 (34.5) | 22.1 (26.8)
  Mirvetuximab Soravtansine: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 53 | 3 | 4 | 8 | 2 | 4 | 7 | 3 | 8 | 40 | 39
  Mirvetuximab Soravtansine: Cycle 3 | NA (NA) — Geometric mean CL could not be calculated for n<3 | 16.9 (34.4) | 17.7 (23) | 16.5 (26.9) | 18.3 (21.4) | 19.3 (17.9) | 18.2 (14) | 17.2 (24.9) | NA (NA) — Geometric mean CL could not be calculated for n<3 | 20.3 (23.9) | 24.3 (21.4) | 26.4 (25) | 18.3 (36.8) | 17.7 (35.6) | 19.2 (23.6)
  Total Antibody: Cycle 1: number analyzed (Participants) | 2 | 7 | 15 | 20 | 50 | 4 | 4 | 9 | 4 | 3 | 6 | 4 | 7 | 31 | 32
  Total Antibody: Cycle 1 | NA (NA) — Geometric mean CL could not be calculated for n<3 | 18 (23.8) | 17.5 (36.5) | 16.7 (33.9) | 16.3 (25.9) | 16.3 (19.8) | 24.5 (24.6) | 16.6 (36.1) | 14.7 (47.1) | 19.3 (83.4) | 15.7 (34.6) | 21.1 (15.2) | 22.6 (49.2) | 20 (44.7) | 16.1 (26.7)
  Total Antibody: Cycle 3: number analyzed (Participants) | 2 | 4 | 10 | 18 | 28 | 2 | 0 | 3 | 2 | 2 | 6 | 2 | 3 | 20 | 17
  Total Antibody: Cycle 3 | NA (NA) — Geometric mean CL could not be calculated for n<3 | 15 (34.3) | 11.7 (27.3) | 11.2 (43.3) | 10.7 (26) | NA (NA) — Geometric mean CL could not be calculated for n<3 |  | 11.1 (20.5) | NA (NA) — Geometric mean CL could not be calculated for n<3 | NA (NA) — Geometric mean CL could not be calculated for n<3 | 13.9 (40.5) | NA (NA) — Geometric mean CL could not be calculated for n<3 | 16.4 (63.9) | 12.9 (57.5) | 9.69 (38.1)

13. Secondary Outcome: PK Parameter: CL of DM4 and SmDM4
Description: as for outcome 12
Time Frame: as for outcome 9
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 2 | 10 | 20 | 32 | 57 | 4 | 4 | 9 | 4 | 4 | 7 | 4 | 10 | 43 | 37
L/h
  DM4: Cycle 1: number analyzed (Participants) | 2 | 10 | 20 | 29 | 54 | 4 | 4 | 9 | 3 | 4 | 5 | 3 | 10 | 43 | 37
  DM4: Cycle 1 | NA (NA) — Geometric mean CL could not be calculated for n<3 | 29 (19.3) | 30.9 (31.5) | 25.2 (36.6) | 28.6 (33.3) | 35 (14.6) | 30.7 (26.8) | 21.8 (64.7) | 25.1 (59.3) | 37.4 (28.3) | 28.2 (52.2) | 35.5 (57.2) | 28.8 (30.7) | 27.7 (27.5) | 29.1 (40.4)
  DM4: Cycle 3: number analyzed (Participants) | 2 | 8 | 15 | 29 | 50 | 3 | 4 | 8 | 1 | 3 | 6 | 3 | 8 | 39 | 36
  DM4: Cycle 3 | NA (NA) — Geometric mean CL could not be calculated for n<3 | 23.5 (26.4) | 28.9 (33) | 22.7 (39.7) | 27.2 (35.5) | 38.6 (16) | 34.5 (23.4) | 22.1 (45.8) | NA (NA) — Geometric mean CL could not be calculated for n<3 | 33.5 (41.5) | 26.6 (54.3) | 44.6 (22.3) | 28.8 (44.4) | 26.7 (31.8) | 29.5 (31.5)
  S-methyl DM4: Cycle 1: number analyzed (Participants) | 2 | 8 | 19 | 32 | 57 | 3 | 2 | 9 | 4 | 4 | 6 | 4 | 9 | 40 | 35
  S-methyl DM4: Cycle 1 | NA (NA) — Geometric mean CL could not be calculated for n<3 | 4.49 (40.2) | 4.77 (61.1) | 3.84 (57.9) | 3.82 (60.8) | 4.39 (52) | NA (NA) — Geometric mean CL could not be calculated for n<3 | 3.35 (70.6) | 3.9 (59.6) | 4.21 (119) | 4.17 (62.8) | 3.42 (73) | 2.78 (91.8) | 3.06 (63.2) | 4.25 (57.1)
  S-methyl DM4: Cycle 3: number analyzed (Participants) | 2 | 10 | 17 | 31 | 50 | 3 | 3 | 8 | 2 | 4 | 7 | 2 | 8 | 38 | 36
  S-methyl DM4: Cycle 3 | NA (NA) — Geometric mean CL could not be calculated for n<3 | 4.18 (66.4) | 4.97 (48.6) | 3.84 (50.5) | 3.87 (52.7) | 5.19 (20.3) | 4.19 (48.3) | 4.26 (59) | NA (NA) — Geometric mean CL could not be calculated for n<3 | 3.9 (83.4) | 3.45 (56.3) | NA (NA) — Geometric mean CL could not be calculated for n<3 | 3.22 (81.9) | 3.57 (63.9) | 4.78 (60.4)

14. Secondary Outcome: PK Parameter: Volume of Distribution at Steady State (Vss) of Mirvetuximab Soravtansine, Total Antibody, DM4, and SmDM4
Description: Blood samples from participants were analyzed to characterize PK when administered in 3- or 4-week cycles.
Time Frame: as for outcome 9
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 3 | 11 | 20 | 34 | 60 | 4 | 4 | 10 | 4 | 5 | 7 | 4 | 10 | 45 | 41
L
  Mirvetuximab Soravtansine Cycle 1: number analyzed (Participants) | 3 | 11 | 20 | 34 | 60 | 4 | 4 | 10 | 4 | 4 | 7 | 4 | 10 | 45 | 41
  Mirvetuximab Soravtansine Cycle 1 | 2.93 (18.2) | 3.63 (12.4) | 3.54 (19.7) | 3.31 (18.5) | 3.87 (25.2) | 3.23 (7.04) | 4.29 (11.9) | 3.52 (23.3) | 3.69 (17.9) | 3.8 (10.7) | 3.88 (24.1) | 4.58 (20.9) | 3.78 (21.8) | 3.59 (23.1) | 3.73 (23)
  Mirvetuximab Soravtansine Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 53 | 3 | 4 | 8 | 2 | 4 | 7 | 3 | 8 | 40 | 39
  Mirvetuximab Soravtansine Cycle 3 | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 3.21 (14.1) | 3.25 (13.2) | 2.83 (23.3) | 3.23 (23.4) | 3.37 (13.3) | 3.4 (15.7) | 3.13 (12.5) | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 3.78 (16.6) | 3.98 (19) | 3.94 (15.4) | 3.28 (31) | 3.1 (25.8) | 3.51 (21.6)
  Total Antibody Cycle 1: number analyzed (Participants) | 2 | 7 | 15 | 20 | 50 | 4 | 4 | 9 | 4 | 3 | 6 | 4 | 7 | 31 | 32
  Total Antibody Cycle 1 | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 4.38 (16.1) | 4.05 (22.7) | 3.9 (34.9) | 4.06 (23.9) | 4.03 (28.1) | 5.67 (10.7) | 4.27 (24.4) | 4.48 (39.2) | 5.01 (1.58) | 4.09 (17.2) | 5.33 (18.7) | 4.69 (23) | 4.09 (30.1) | 4.21 (25.6)
  Total Antibody Cycle 3: number analyzed (Participants) | 2 | 4 | 10 | 18 | 28 | 2 | 0 | 3 | 2 | 2 | 6 | 2 | 3 | 20 | 17
  Total Antibody Cycle 3 | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 3.74 (23.7) | 3.17 (17.2) | 2.97 (34.6) | 2.95 (24.4) | NA (NA) — Geometric mean Vss could not be calculated for n<3 |  | 3.09 (8.55) | NA (NA) — Geometric mean Vss could not be calculated for n<3 | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 3.76 (49.6) | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 4.01 (57.5) | 3.28 (30.5) | 2.9 (25.4)
  DM4 Cycle 1: number analyzed (Participants) | 2 | 10 | 20 | 29 | 54 | 4 | 4 | 9 | 3 | 4 | 5 | 3 | 10 | 43 | 37
  DM4 Cycle 1 | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 2590 (23.8) | 2490 (31.4) | 2010 (38.6) | 2240 (40.4) | 2670 (20.9) | 2580 (59.4) | 1720 (36) | 1880 (51.6) | 2730 (26.5) | 2010 (53.5) | 2100 (80.9) | 2410 (52.5) | 2060 (31.1) | 2350 (45.1)
  DM4 Cycle 3: number analyzed (Participants) | 2 | 8 | 15 | 29 | 50 | 3 | 4 | 8 | 1 | 3 | 6 | 3 | 8 | 39 | 36
  DM4 Cycle 3 | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 2190 (20.7) | 2480 (24.3) | 1990 (43.7) | 2370 (35.9) | 3030 (7.84) | 3160 (7.05) | 1900 (55.6) | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 3300 (38.4) | 2140 (35.9) | 2930 (22.9) | 2450 (53.6) | 2270 (32.8) | 2450 (29.1)
  SmDM4 Cycle 1: number analyzed (Participants) | 2 | 8 | 19 | 32 | 57 | 3 | 2 | 9 | 4 | 4 | 6 | 4 | 9 | 40 | 35
  SmDM4 Cycle 1 | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 911 (57.3) | 900 (67.1) | 731 (69.3) | 751 (66.7) | 932 (63.7) | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 652 (65) | 832 (61.6) | 1100 (114) | 855 (66.3) | 695 (81.2) | 547 (97.6) | 592 (66.4) | 840 (65.1)
  SmDM4 Cycle 3: number analyzed (Participants) | 2 | 10 | 17 | 31 | 50 | 3 | 3 | 8 | 2 | 4 | 7 | 2 | 8 | 38 | 36
  SmDM4 Cycle 3 | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 761 (53.6) | 878 (48.6) | 698 (51.8) | 696 (51) | 1100 (1.87) | 833 (24.5) | 754 (60.7) | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 947 (82.5) | 773 (64.7) | NA (NA) — Geometric mean Vss could not be calculated for n<3 | 621 (76.2) | 709 (59.1) | 891 (67.2)

15. Secondary Outcome: PK Parameter: Time to Reach Cmax (Tmax) of Mirvetuximab Soravtansine, Total Antibody, DM4, and SmDM4
Description: Blood samples from participants were analyzed to characterize the PK of mirvetuximab soravtansine when administered in 3- or 4-week cycles.
  PK parameters were derived using non-compartmental PK analysis.
Time Frame: as for outcome 11
Population: as for outcome 7
Measure: Median (Full Range); unit: h
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Regimen D Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen D Dose Expansion: Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 3 | 11 | 20 | 35 | 60 | 4 | 4 | 10 | 4 | 5 | 7 | 4 | 10 | 46 | 41
h
  Mirvetuximab Soravtansine: Cycle 1 | 1.75 [1.52 to 1.85] | 1.9 [1.32 to 7.48] | 2.1 [1.63 to 7.8] | 1.92 [1.62 to 8.08] | 2.06 [1.42 to 24] | 1.68 [1.63 to 1.72] | 1.96 [1.72 to 7.78] | 1.86 [1.5 to 7.57] | 4.28 [1.22 to 7.62] | 1.73 [1.45 to 7.08] | 5.98 [1.73 to 8.05] | 2 [1.67 to 7.57] | 2.14 [1.87 to 7.72] | 2.12 [1.62 to 8.23] | 2.07 [1.47 to 8.22]
  Mirvetuximab Soravtansine: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 58 | 4 | 4 | 9 | 2 | 4 | 7 | 3 | 8 | 41 | 41
  Mirvetuximab Soravtansine: Cycle 3 | NA [NA to NA] — As per the PK analysis plan, Tmax statistics were not calculated when less than 3 individual values were available. | 3.88 [0.967 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported. | 3.46 [1.17 to 7.5] | 2.24 [1.02 to 7.37] | 1.49 [1.08 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported. | 4.06 [0.95 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported. | 1.02 [0.95 to 5.35] | 1.48 [1.07 to 5.97] | NA [NA to NA] — As per the PK analysis plan, Tmax statistics were not calculated when less than 3 individual values were available. | 4.04 [1.2 to 7] | 6.08 [1.15 to 7.33] | 1.45 [1.17 to 22] | 1.26 [1.15 to 7.1] | 1.5 [0.95 to 25.6] | 6.98 [0.95 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported.
  Total Antibody: Cycle 1 | 1.75 [1.52 to 5.52] | 1.9 [1.32 to 7.75] | 2.1 [1.63 to 25.6] | 1.9 [1.62 to 48.2] | 2.05 [1.48 to 9] | 1.68 [1.63 to 24.1] | 4.09 [1.72 to 7.78] | 1.88 [1.5 to 7.55] | 3.84 [1.63 to 6.75] | 1.87 [1.45 to 7.53] | 5.98 [1.67 to 25] | 4.82 [1.67 to 7.87] | 2.25 [1.88 to 48.9] | 2.08 [1.43 to 8.05] | 2.2 [1.13 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported.
  Total Antibody: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 58 | 4 | 4 | 9 | 2 | 4 | 7 | 3 | 8 | 41 | 41
  Total Antibody: Cycle 3 | NA [NA to NA] — As per the PK analysis plan, Tmax statistics were not calculated when less than 3 individual values were available. | 3.88 [0.967 to 48.9] | 3.68 [1.08 to 25.2] | 2.24 [1.02 to 27.2] | 1.49 [1.08 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported. | 6.91 [1.02 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported. | 1.03 [0.95 to 7.05] | 1.48 [1.17 to 5.83] | NA [NA to NA] — As per the PK analysis plan, Tmax statistics were not calculated when less than 3 individual values were available. | 1.23 [1.05 to 6.83] | 7.12 [6.08 to 49.6] | 7.1 [1.05 to 48.7] | 3.7 [1.15 to 24] | 1.63 [0.95 to 25.1] | 3.03 [0.967 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported.
  DM4: Cycle 1 | 7.2 [5.52 to 7.27] | 7.5 [1.32 to 26.4] | 7.78 [1.83 to 8.58] | 7.63 [0 to 22.4] | 7.58 [1.67 to 24] | 7.4 [1.72 to 7.6] | 7.56 [6 to 7.78] | 7.34 [5.87 to 21.5] | 7.12 [5.87 to 7.62] | 7.32 [6 to 7.53] | 5.98 [1.67 to 8.05] | 7.62 [7.53 to 7.87] | 7.7 [2.25 to 8.22] | 7.58 [1.73 to 24] | 7.67 [1.58 to 8.22]
  DM4: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 58 | 4 | 4 | 9 | 2 | 4 | 7 | 3 | 8 | 41 | 41
  DM4: Cycle 3 | NA [NA to NA] — As per the PK analysis plan, Tmax statistics were not calculated when less than 3 individual values were available. | 7 [1.25 to 7.75] | 7.06 [1.25 to 7.63] | 6.94 [1.08 to 7.82] | 6.96 [1.1 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported. | 6.99 [6.82 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported. | 6.96 [5.35 to 7.05] | 6.08 [5.03 to 7.77] | NA [NA to NA] — As per the PK analysis plan, Tmax statistics were not calculated when less than 3 individual values were available. | 6.89 [1.2 to 7] | 7.02 [6.08 to 7.33] | 7.1 [1.05 to 7.6] | 7.08 [1.33 to 7.45] | 7.03 [0.95 to 24.8] | 7.13 [0.95 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported.
  S-methyl DM4: Cycle 1 | 23.8 [7.2 to 119] | 23.9 [5.87 to 170] | 7.83 [5.87 to 46.7] | 7.83 [5.68 to 166] | 8.26 [6.05 to 170] | 48.2 [24.6 to 169] | 108 [25.4 to 170] | 7.34 [5.87 to 163] | 23.8 [6.75 to 23.9] | 23.8 [7.53 to 24.4] | 7.7 [5.98 to 50.4] | 7.72 [7.53 to 49.6] | 7.84 [6.17 to 167] | 8 [7.18 to 171] | 8.15 [6.93 to 167]
  S-methyl DM4: Cycle 3: number analyzed (Participants) | 2 | 10 | 18 | 32 | 58 | 4 | 4 | 9 | 2 | 4 | 7 | 3 | 8 | 41 | 41
  S-methyl DM4: Cycle 3 | NA [NA to NA] — As per the PK analysis plan, Tmax statistics were not calculated when less than 3 individual values were available. | 7.01 [5.83 to 24.6] | 7.17 [5.83 to 47.7] | 7.11 [5.67 to 48.7] | 7.41 [6.02 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported. | 6.99 [6.82 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported. | 15.1 [5.35 to 47.6] | 6.08 [5.03 to 21.3] | NA [NA to NA] — As per the PK analysis plan, Tmax statistics were not calculated when less than 3 individual values were available. | 7.04 [6.83 to 47.2] | 7.02 [6.08 to 7.33] | 7.1 [6.87 to 7.6] | 7.08 [6.08 to 7.45] | 7.12 [0.95 to 47.3] | 7.22 [0.95 to NA] — NA = Insufficient number of participants with events (data samples) for accurate calculation of Tmax upper range, therefore, not reported.

16. Secondary Outcome: Plasma Concentration of Bevacizumab
Description: Blood samples from participants at the end of infusion were analyzed to characterize the PK of mirvetuximab soravtansine when administered in 3- or 4-week cycles.
Time Frame: At end of infusion (EOI) of Cycle 1; and at pre-infusion and EOI of Cycles 2 to 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Regimen A Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Regimen A Dose Expansion Cohort 1: Bevacizumab-naïve | Regimen A Dose Expansion Cohort 2: Bevacizumab Pre-treated | Regimen A Dose Expansion Cohort 3: Pt-agnostic: | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 3 | 11 | 20 | 33 | 59 | 40
ug/mL
  Cycle 1 EOI: number analyzed (Participants) | 3 | 11 | 20 | 33 | 59 | 38
  Cycle 1 EOI | 368 (20.2) | 352 (31.9) | 406 (22.3) | 430 (19.3) | 448 (23.2) | 413 (23.9)
  Cycle 2 Pre-infusion: number analyzed (Participants) | 3 | 11 | 19 | 32 | 59 | 39
  Cycle 2 Pre-infusion | 69.3 (37) | 66 (35.4) | 90.6 (57.8) | 87.5 (37.4) | 88.1 (35) | 92.5 (39.9)
  Cycle 2 EOI: number analyzed (Participants) | 3 | 8 | 20 | 31 | 54 | 39
  Cycle 2 EOI | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 477 (23.8) | 429 (38.2) | 528 (20.8) | 559 (28.4) | 473 (44.6)
  Cycle 3 Pre-infusion: number analyzed (Participants) | 2 | 9 | 18 | 31 | 54 | 37
  Cycle 3 Pre-infusion | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 79.9 (52.9) | 132 (17) | 117 (39.3) | 118 (51.2) | 127 (45.8)
  Cycle 3 EOI: number analyzed (Participants) | 2 | 10 | 16 | 31 | 51 | 38
  Cycle 3 EOI | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 408 (59.2) | 540 (23.6) | 556 (17.8) | 616 (22.1) | 531 (33.1)
  Cycle 4 Pre-infusion: number analyzed (Participants) | 2 | 8 | 17 | 28 | 51 | 38
  Cycle 4 Pre-infusion | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 133 (24.1) | 134 (51.1) | 141 (49.4) | 123 (78.2) | 132 (92.9)
  Cycle 4 EOI: number analyzed (Participants) | 2 | 10 | 17 | 30 | 46 | 40
  Cycle 4 EOI | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 537 (25.2) | 539 (20.7) | 505 (39.1) | 584 (35.7) | 485 (128)
  Cycle 5 Pre-infusion: number analyzed (Participants) | 2 | 5 | 16 | 25 | 44 | 37
  Cycle 5 Pre-infusion | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 134 (18.3) | 163 (28.9) | 151 (36.1) | 137 (61) | 153 (51)
  Cycle 5 EOI: number analyzed (Participants) | 2 | 6 | 16 | 25 | 43 | 37
  Cycle 5 EOI | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 583 (31.1) | 565 (19.1) | 587 (20.3) | 558 (80.6) | 547 (24.1)
  Cycle 6 Pre-infusion: number analyzed (Participants) | 2 | 5 | 12 | 24 | 41 | 39
  Cycle 6 Pre-infusion | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 80.7 (96.8) | 191 (27.6) | 149 (37.8) | 166 (29.6) | 170 (51.5)
  Cycle 6 EOI: number analyzed (Participants) | 1 | 7 | 12 | 23 | 38 | 38
  Cycle 6 EOI | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 513 (29.1) | 574 (26.2) | 559 (23.9) | 654 (24.6) | 525 (39.8)

17. Secondary Outcome: Plasma Concentration of Carboplatin
Description: as for outcome 16
Time Frame: At end of infusion, 6 and 24 hours post-infusion of Cycle 1; and at pre-infusion and end of infusion of Cycles 2, 4, 5 and 6; at pre-infusion, end of infusion and 6 and 24 hours post-infusion of Cycle 3
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Regimen B Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Regimen E: Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
Number analyzed (Participants) | 4 | 4 | 9 | 41
ng/mL
  Cycle 1: EOI: number analyzed (Participants) | 4 | 4 | 9 | 37
  Cycle 1: EOI | 10300 (11.3) | 1060 (35.2) | 13900 (19) | 11800 (25.6)
  Cycle 1: 6 hours post-infusion: number analyzed (Participants) | 4 | 4 | 9 | 0
  Cycle 1: 6 hours post-infusion | 2890 (45.6) | 3790 (10.3) | 3120 (151) |
  Cycle 1 24 hours post-infusion: number analyzed (Participants) | 3 | 4 | 9 | 36
  Cycle 1 24 hours post-infusion | 719 (4.77) | 913 (19.7) | 1030 (43.8) | 817 (35)
  Cycle 2: Pre-infusion: number analyzed (Participants) | 4 | 3 | 6 | 38
  Cycle 2: Pre-infusion | 124 (14.8) | 142 (21.7) | 158 (13.5) | 170 (79.2)
  Cycle 2: EOI: number analyzed (Participants) | 3 | 4 | 9 | 40
  Cycle 2: EOI | 10800 (22) | 11600 (18.5) | 11700 (80.9) | 11000 (146)
  Cycle 3: Pre-infusion: number analyzed (Participants) | 2 | 3 | 6 | 40
  Cycle 3: Pre-infusion | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 245 (34.6) | 173 (35.9) | 203 (28.2)
  Cycle 3: EOI: number analyzed (Participants) | 2 | 4 | 8 | 41
  Cycle 3: EOI | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 4170 (946) | 12100 (28.9) | 12300 (26.9)
  Cycle 3: 6 hours post-infusion: number analyzed (Participants) | 3 | 4 | 8 | 0
  Cycle 3: 6 hours post-infusion | 1140 (412) | 3890 (29.9) | 1630 (238) |
  Cycle 3: 24 hours post-infusion: number analyzed (Participants) | 2 | 4 | 7 | 35
  Cycle 3: 24 hours post-infusion | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 1330 (27.3) | 1270 (41.3) | 1440 (49)
  Cycle 4: Pre-infusion: number analyzed (Participants) | 3 | 3 | 6 | 36
  Cycle 4: Pre-infusion | 220 (31.8) | 243 (59.1) | 214 (20.6) | 250 (39.9)
  Cycle 4: EOI: number analyzed (Participants) | 3 | 2 | 8 | 38
  Cycle 4: EOI | 8230 (43.9) | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 214 (20.6) | 12500 (29.9)
  Cycle 5: Pre-infusion: number analyzed (Participants) | 3 | 2 | 6 | 35
  Cycle 5: Pre-infusion | 199 (41.8) | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 194 (37.9) | 270 (43)
  Cycle 5: EOI: number analyzed (Participants) | 3 | 2 | 8 | 36
  Cycle 5: EOI | 10900 (36.9) | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 13800 (31.8) | 11200 (88.1)
  Cycle 6: Pre-infusion: number analyzed (Participants) | 3 | 2 | 8 | 37
  Cycle 6: Pre-infusion | 251 (20.2) | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 234 (24.6) | 271 (45.4)
  Cycle 6: EOI: number analyzed (Participants) | 3 | 2 | 8 | 35
  Cycle 6: EOI | 12100 (32.5) | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 12100 (32.1) | 10700 (77.9)

18. Secondary Outcome: Plasma Concentration of Pegylated Liposomal Doxorubicin
Description: as for outcome 16
Time Frame: At end of infusion of Cycle 1; and at pre-infusion and end of infusion of Cycles 2 to 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Regimen C Dose Escalation: Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2
Number analyzed (Participants) | 4 | 5 | 7
ng/mL
  Cycle 1: EOI: number analyzed (Participants) | 4 | 5 | 5
  Cycle 1: EOI | 18700 (8.72) | 24400 (14.3) | 26400 (7.85)
  Cycle 2: Pre-infusion: number analyzed (Participants) | 0 | 1 | 5
  Cycle 2: Pre-infusion |  | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 226 (44.9)
  Cycle 2: EOI: number analyzed (Participants) | 4 | 3 | 7
  Cycle 2: EOI | 17300 (17.1) | 25700 (6.88) | 26100 (12.1)
  Cycle 3: Pre-infusion: number analyzed (Participants) | 1 | 4 | 5
  Cycle 3: Pre-infusion | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 228 (63)
  Cycle 3: EOI: number analyzed (Participants) | 2 | 4 | 7
  Cycle 3: EOI | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 26200 (12.8) | 26200 (14.3)
  Cycle 4: Pre-infusion: number analyzed (Participants) | 0 | 1 | 5
  Cycle 4: Pre-infusion |  | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 151 (54.2)
  Cycle 4: EOI: number analyzed (Participants) | 2 | 3 | 7
  Cycle 4: EOI | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 24300 (24.1) | 24400 (15.4)
  Cycle 5: Pre-infusion: number analyzed (Participants) | 0 | 1 | 5
  Cycle 5: Pre-infusion |  | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 177 (81.1)
  Cycle 5: EOI: number analyzed (Participants) | 2 | 4 | 7
  Cycle 5: EOI | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 23700 (17.1) | 25000 (11.3)
  Cycle 6: Pre-infusion: number analyzed (Participants) | 0 | 1 | 5
  Cycle 6: Pre-infusion |  | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 157 (134)
  Cycle 6: EOI: number analyzed (Participants) | 1 | 3 | 7
  Cycle 6: EOI | NA (NA) — Geometric mean plasma concentration could not be calculated for n<3 | 22900 (13.3) | 24600 (14.7)

19. Secondary Outcome: Immunogenicity: Number of Participants With Anti-Drug Antibody (ADA) Response to Mirvetuximab Soravtansine
Description: Blood samples were collected to measure the presence of ADAs for mirvetuximab soravtansine. Seronegative is defined as a participant that tests negative at all visits. Treatment-emergent ADA is defined as a participant that is seronegative prior to dosing on Day 1 of Cycle 1 and tests positive in both screening and confirmatory assays at one or more subsequent visits. Treatment-unaffected ADA is defined as a participant test positive in both screening and confirmatory assays prior to dosing on Day 1 of Cycle 1 with a post-dose titer increase of less than or equal to 4-fold (based on a 2-fold sample dilution). Treatment-boosted ADA is defined as a participant test positive in both screening and confirmatory assays prior to dosing on Day 1 of Cycle 1 with a post-dose titer increase of more than a 4-fold increase (based on a 2-fold sample dilution).
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (maximum exposure: 283.3 weeks)
Population: The immunogenicity population included all participants who received at least 1 dose of study drug and have evaluable immunogenicity data. As per analysis plan, all regimens (arms/groups) were combined for each phase of the study (dose escalation and dose expansion) for analysis of ADA.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation Phase: All participants who received mirvetuximab soravtansine during the dose escalation phase of the study (Regimens A, B, C, and D).
- Dose Expansion Phase: All participants who received mirvetuximab soravtansine during the dose expansion phase of the study (Regimens A, D, and E).
Arm/Group | Dose Escalation Phase | Dose Expansion Phase
Number analyzed (Participants) | 62 | 202
Participants
  Seronegative | 51 | 175
  Treatment-emergent ADA | 3 | 11
  Treatment-unaffected ADA | 7 | 11
  Treatment-boosted ADA | 1 | 5

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (maximum exposure: 238.3 weeks)
Description: Safety population included all participants who were enrolled and received at least 1 dose of study drug. AEs (serious and non-serious) and deaths occurred during TEAE period were reported. Data were reported by dose group and where applicable the dose-escalation and expansion phases were combined to report data by dose group.
Groups:
- Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2: Participants were administered mirvetuximab soravtansine 5 mg/kg + PLD 40 mg/m^2 on Day 1 of each 28-day cycle.
Arm/Group | Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg | Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg | Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 | Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 | Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 | Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 | Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 | Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 | Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg | Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg | Mirvetuximab Soravtansine + Bevacizumab + Carboplatin
All-Cause Mortality (participants affected / at risk) | 0/3 | 5/126 | 0/4 | 0/4 | 0/10 | 0/4 | 0/5 | 0/7 | 0/4 | 4/56 | 2/41
Serious Adverse Events (participants affected / at risk) | 2/3 | 49/126 | 2/4 | 4/4 | 3/10 | 1/4 | 2/5 | 3/7 | 2/4 | 25/56 | 17/41
Other Adverse Events (participants affected / at risk) | 3/3 | 125/126 | 4/4 | 4/4 | 10/10 | 4/4 | 4/5 | 7/7 | 4/4 | 56/56 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg (N=3) | Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg (N=126) | Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 (N=4) | Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 (N=4) | Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 (N=10) | Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 (N=4) | Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 (N=5) | Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 (N=7) | Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg (N=4) | Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg (N=56) | Mirvetuximab Soravtansine + Bevacizumab + Carboplatin (N=41)
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 7 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Colitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric varices (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Sepsis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device malfunction (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraneoplastic dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
IgA nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirvetuximab Soravtansine 5 mg/kg + Bevacizumab 15 mg/kg (N=3) | Mirvetuximab Soravtansine 6 mg/kg + Bevacizumab 15 mg/kg (N=126) | Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC4 (N=4) | Mirvetuximab Soravtansine 5 mg/kg + Carboplatin AUC5 (N=4) | Mirvetuximab Soravtansine 6 mg/kg + Carboplatin AUC5 (N=10) | Mirvetuximab Soravtansine 5 mg/kg + PLD 30 mg/m^2 (N=4) | Mirvetuximab Soravtansine 5 mg/kg + PLD 40 mg/m^2 (N=5) | Mirvetuximab Soravtansine 6 mg/kg + PLD 40 mg/m^2 (N=7) | Mirvetuximab Soravtansine 5 mg/kg + Pembrolizumab 200 mg (N=4) | Mirvetuximab Soravtansine 6 mg/kg + Pembrolizumab 200 mg (N=56) | Mirvetuximab Soravtansine + Bevacizumab + Carboplatin (N=41)
Diarrhoea (Gastrointestinal disorders) | 1 | 85 | 4 | 3 | 5 | 3 | 4 | 4 | 2 | 32 | 34
Nausea (Gastrointestinal disorders) | 2 | 73 | 1 | 2 | 10 | 1 | 4 | 6 | 3 | 30 | 33
Vomiting (Gastrointestinal disorders) | 2 | 45 | 2 | 1 | 6 | 1 | 3 | 3 | 2 | 20 | 21
Abdominal pain (Gastrointestinal disorders) | 1 | 44 | 0 | 0 | 2 | 1 | 2 | 2 | 0 | 18 | 23
Abdominal distension (Gastrointestinal disorders) | 1 | 33 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 9 | 10
Constipation (Gastrointestinal disorders) | 1 | 33 | 0 | 1 | 4 | 2 | 4 | 2 | 2 | 16 | 12
Abdominal pain upper (Gastrointestinal disorders) | 0 | 18 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 9 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 14 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 8 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 13 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 8 | 5
Stomatitis (Gastrointestinal disorders) | 1 | 12 | 1 | 0 | 0 | 0 | 1 | 4 | 0 | 3 | 7
Ascites (Gastrointestinal disorders) | 0 | 10 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 6 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 6 | 6
Colitis (Gastrointestinal disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Frequent bowel movements (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyschezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal mucosa hyperaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival recession (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Oral mucosal hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Teeth brittle (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 67 | 2 | 2 | 7 | 1 | 4 | 4 | 4 | 28 | 30
Asthenia (General disorders) | 0 | 24 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4
Pyrexia (General disorders) | 0 | 18 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 5 | 4
Early satiety (General disorders) | 0 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Oedema peripheral (General disorders) | 0 | 11 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 6 | 7
Chills (General disorders) | 0 | 9 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 2
Non-cardiac chest pain (General disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Pain (General disorders) | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Catheter site pain (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Gait disturbance (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Mucosal inflammation (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Administration site extravasation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site discolouration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site injury (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pruritus (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Extravasation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Implant site dehiscence (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3
Pelvic mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sense of oppression (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Medical device site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Physical deconditioning (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaccination site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaccination site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaccination site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 32 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 14 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 29 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 25 | 1 | 3 | 4 | 0 | 2 | 3 | 0 | 12 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 24 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 9
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 18 | 1 | 2 | 2 | 0 | 0 | 1 | 0 | 11 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 12 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 12 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 43 | 1 | 1 | 3 | 0 | 3 | 2 | 0 | 12 | 23
Neuropathy peripheral (Nervous system disorders) | 1 | 33 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 15 | 14
Dysgeusia (Nervous system disorders) | 0 | 17 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 5 | 8
Dizziness (Nervous system disorders) | 0 | 15 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 8 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 14 | 0 | 1 | 6 | 0 | 0 | 2 | 2 | 15 | 7
Neurotoxicity (Nervous system disorders) | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Amnesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgraphia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Resting tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial spasm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 2 | 71 | 3 | 3 | 6 | 0 | 3 | 3 | 2 | 26 | 31
Dry eye (Eye disorders) | 1 | 39 | 0 | 1 | 4 | 0 | 1 | 2 | 1 | 20 | 16
Keratopathy (Eye disorders) | 0 | 37 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 10 | 20
Cataract (Eye disorders) | 1 | 25 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 6 | 11
Visual acuity reduced (Eye disorders) | 0 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 8
Photophobia (Eye disorders) | 0 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5
Eye pain (Eye disorders) | 0 | 13 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 9 | 7
Corneal cyst (Eye disorders) | 0 | 8 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2
Diplopia (Eye disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4
Foreign body sensation in eyes (Eye disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 1 | 4 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 0
Vitreous floaters (Eye disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4
Corneal deposits (Eye disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Visual impairment (Eye disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Glaucoma (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angle closure glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphakia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal epithelium defect (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corneal toxicity (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye allergy (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glare (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Meibomian gland dysfunction (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Optic atrophy (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Optic disc drusen (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pinguecula (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pterygium (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous opacities (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acquired corneal dystrophy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blindness transient (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corneal epithelial microcysts (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lenticular opacities (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Maculopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meibomianitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orbital oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Posterior capsule opacification (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal drusen (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Trichiasis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 47 | 0 | 3 | 3 | 0 | 0 | 3 | 2 | 15 | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 27 | 4 | 1 | 2 | 0 | 0 | 0 | 1 | 6 | 9
Dehydration (Metabolism and nutrition disorders) | 1 | 21 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 13 | 3 | 2 | 3 | 2 | 0 | 3 | 1 | 12 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 8 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 26 | 1 | 1 | 3 | 0 | 0 | 1 | 0 | 12 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 24 | 0 | 0 | 5 | 0 | 1 | 1 | 0 | 13 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 20 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 9 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 17 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 6 | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 16 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 13 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 6 | 7
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enthesophyte (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 34 | 0 | 2 | 3 | 0 | 2 | 3 | 0 | 21 | 13
Weight decreased (Investigations) | 1 | 32 | 0 | 0 | 2 | 1 | 1 | 3 | 0 | 8 | 11
Alanine aminotransferase increased (Investigations) | 0 | 31 | 0 | 2 | 3 | 0 | 1 | 3 | 0 | 19 | 10
Blood alkaline phosphatase increased (Investigations) | 0 | 13 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 7 | 2
Blood creatinine increased (Investigations) | 0 | 3 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 6 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Albumin urine present (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ammonia increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial test (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 29 | 1 | 0 | 2 | 2 | 2 | 2 | 0 | 9 | 12
Nasopharyngitis (Infections and infestations) | 0 | 13 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4
Sinusitis (Infections and infestations) | 0 | 9 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 9 | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 5 | 4
Pneumonia (Infections and infestations) | 0 | 6 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 4 | 1
Oral herpes (Infections and infestations) | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess jaw (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Clitoris abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail bed infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyuria (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Corneal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Keratitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmic herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papilloma viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 41 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 4 | 15
Flushing (Vascular disorders) | 0 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 4
Hot flush (Vascular disorders) | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Hypotension (Vascular disorders) | 0 | 5 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 37 | 2 | 3 | 6 | 0 | 1 | 2 | 0 | 4 | 29
Neutropenia (Blood and lymphatic system disorders) | 0 | 23 | 1 | 2 | 7 | 0 | 3 | 2 | 0 | 1 | 21
Anaemia (Blood and lymphatic system disorders) | 0 | 11 | 0 | 2 | 5 | 2 | 0 | 3 | 1 | 9 | 13
Leukopenia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Acquired porokeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic pigmented purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spider naevus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin fragility (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 18 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 10 | 6
Anxiety (Psychiatric disorders) | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 7
Confusional state (Psychiatric disorders) | 0 | 6 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 5 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 5
Agitation (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
Dysuria (Renal and urinary disorders) | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Micturition urgency (Renal and urinary disorders) | 0 | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder discomfort (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 6
Fall (Injury, poisoning and procedural complications) | 2 | 7 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 3 | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 4 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulva cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulval haematoma (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Deafness (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ototoxicity (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Tachycardia (Cardiac disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contrast media reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Device occlusion (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corrective lens user (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraocular lens implant (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal affective disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acquired corneal dystrophy (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meibomian gland dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT02606305/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT02606305/SAP_001.pdf